CLINICAL TRIAL: NCT04664010
Title: Efficacy and Safety of High-dose Vitamin C Combined With Traditional Chinese Medicine in the Treatment of Moderate and Severe Coronavirus Pneumonia (COVID-19)
Brief Title: Efficacy and Safety of High-dose Vitamin C Combined With Chinese Medicine Against Coronavirus Pneumonia (COVID-19)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an International Medical Center Hospital (Other)
Responsible Party: Principal Investigator, Qiang Yin, President, Xi'an International Medical Center Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XianInternationalMCH_HXJ
Record Dates: First submitted 2020-12-07; First posted 2020-12-11 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
Keywords: COVID-19; vitamin C; traditional Chinese medicine
MeSH Terms: conditions — COVID-19 | interventions — Interferon-alpha; abidol; Ribavirin; Fumigation; Glucose

STUDY DESIGN:
Intervention Model Description: participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: Blinding and blinding maintenance
  (1)The biostatisticians and the personnel unrelated to the clinical trial complete the binding of the study drugs and emergency card preparation. The random coding table and corresponding parameters are recorded blindly. After drug designation, the personnel responsible for blinding of the study drugs will sign at the perforation of the blinding envelope.
  A two-level blinding design will be adopted. The first-level code corresponds to intervention A or intervention B, and the second-level code presents the corresponding group. The envelope containing two-level blinding file will be preserved in Tianjin Angsai Cell Gene Engineering Co., Ltd., China until unblinding. The unblinding will not be performed during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- moderate COVID-19 group (Experimental): patients with moderate COVID-19 receiving western medicine treatment
  Interventions: Drug: Alpha-interferon alpha, abidol, ribavirin, Buzhong Yiqi plus and minus formula, Huhuang Detoxicity Paste, Baimu Qingre Jiedu Paste, fumigation/inhalation of vitamin C
- severe COVID-19 group (Experimental): patients with severe COVID-19 receiving western medicine treatment
  Interventions: Drug: Alpha-interferon alpha, abidol, ribavirin, Buzhong Yiqi plus and minus formula, Huhuang Detoxicity Paste, Baimu Qingre Jiedu Paste, fumigation/inhalation of vitamin C
- moderate COVID-19 with traditional Chinese medicine group (Experimental): patients with moderate COVID-19 receiving western medicine treatment + traditional Chinese medicine + intravenous administration of 5% glucose
  Interventions: Drug: Alpha-interferon, abidol, ribavirin, Buzhong Yiqi plus and minus formula, Huhuang Detoxicity Paste, Baimu Qingre Jiedu Paste and 5% glucose
- moderate COVID-19 with combination therapy group (Experimental): patients with moderate COVID-19 receiving western medicine treatment + traditional Chinese medicine + intravenous administration of 5% glucose containing high-dose vitamin C
  Interventions: Drug: Alpha-interferon, abidol, ribavirin, Buzhong Yiqi plus and minus formula, Huhuang Detoxicity Paste, Baimu Qingre Jiedu Paste and 5% glucose
- severe COVID-19 with traditional Chinese medicine group (Experimental): patients with severe COVID-19 receiving western medicine treatment + traditional Chinese medicine + intravenous administration of 5% glucose
  Interventions: Drug: Alpha-interferon, abidol, ribavirin, Buzhong Yiqi plus and minus formula, Huhuang Detoxicity Paste, Baimu Qingre Jiedu Paste and high-dose vitamin C treatment
- severe COVID-19 with combination therapy group (Experimental): patients with severe COVID-19 receiving western medicine treatment + traditional Chinese medicine + intravenous administration of 5% glucose containing high-dose vitamin C
  Interventions: Drug: Alpha-interferon, abidol, ribavirin, Buzhong Yiqi plus and minus formula, Huhuang Detoxicity Paste, Baimu Qingre Jiedu Paste and high-dose vitamin C treatment

INTERVENTIONS:
Drug: Alpha-interferon alpha, abidol, ribavirin, Buzhong Yiqi plus and minus formula, Huhuang Detoxicity Paste, Baimu Qingre Jiedu Paste, fumigation/inhalation of vitamin C — Atomized inhalation of 5 million U α-interferon and 2 mL sterilized water, twice a day; 0.2 g arbidol, three times a day, treatment course no more than 10 days; intravenous administration of ribavirin 500 mg, once every 12 hours, treatment course no more than 10 days; intravenous administration of 10 g immunoglobulin C, once a day, 3-5 days. Anti-bacterial infection treatment is given to the patients who have yellow sputum and increased levels of procalcitonin and other bacterial infection specific indicators.
  Other Names: Western medicine treatment
  Arms: moderate COVID-19 group; severe COVID-19 group
Drug: Alpha-interferon, abidol, ribavirin, Buzhong Yiqi plus and minus formula, Huhuang Detoxicity Paste, Baimu Qingre Jiedu Paste and 5% glucose — Buzhong Yiqi plus and minus formula: 1 dose once, twice a day, taking with warm water. Huhuang Detoxicity Paste: One dose once, twice a day, taking with warm water; Baimu Qingre Jiedu Paste: One dose once, twice a day, taking with warm water; Fumigation/inhalation of Chinese herbs and vitamin C: 30-40 minutes once, 3-7 times a day. Patients take vitamin E capsule and folic acid every day. plus invention 1
  Other Names: Traditional Chinese medicine treatment plus Western medicine treatment
  Arms: moderate COVID-19 with combination therapy group; moderate COVID-19 with traditional Chinese medicine group
Drug: Alpha-interferon, abidol, ribavirin, Buzhong Yiqi plus and minus formula, Huhuang Detoxicity Paste, Baimu Qingre Jiedu Paste and high-dose vitamin C treatment — invention 1 plus invention 2 plus 100 mL of 5% glucose containing vitamin C (10 g/60 kg body mass) is intravenously administered twice a day.
  Other Names: Traditional Chinese medicine treatment plus Western medicine treatment plus Bolus administration of vitamin C
  Arms: severe COVID-19 with combination therapy group; severe COVID-19 with traditional Chinese medicine group

SUMMARY:
In December 2019, coronavirus pneumonia (COVID-19) was detected in many cases in Wuhan, China. With the rapid spread of the coronavirus, cases of COVID-19 were also reported in other cities of China and other countries. COVID-19 can cause amplification of the pulmonary inflammatory responses, including the production of a large amount of free radicals and the release of inflammatory factors, in a short time after infection, leading to lung tissue damage and dysfunction, even resulting in life-threatening respiratory distress syndrome and respiratory failure. At present, there are no effective drugs targeting COVID-19. Previous studies have shown that Buzhong Yiqi Decoction has anti-bacterial, anti-viral, and anti-allergy effects. High-dose vitamin C also has anti-oxidative and anti-toxin effects, possibly exhibiting good effects in the treatment of viral infection and critical respiratory diseases. The study objectives include (1) investigate whether Buzhong Yiqi Decoction can improve the clinical symptoms of patients with mild and severe COVID-19 and accelerate recovery and to further investigate the clinical efficacy of high-dose vitamin C combined with traditional Chinese medicine in the treatment of mild and severe COVID-19; (2) to assess the safety of high-dose vitamin C combined with Chinese medicine in the treatment of mild and severe COVID-19.

DETAILED DESCRIPTION:
Preparation prior to treatment

1. Record of age, sex, race, height, body mass, body mass index, body temperature, blood pressure, pulse, and respiratory rate;
2. Record of previous medical history, current medical history, treatment history, concomitant disease/treatment history;
3. Record of laboratory tests: routine blood test, routine stool and urine tests, fecal occult blood test, C-reactive protein measurement, biochemical assay, PCR testing for respiratory virus, tumor marker test, and ABO typing
4. Cytokine detection: Serum levels of interleukin-6, interleukin-10, and tumor necrosis factor-alpha (TNF-α)
5. Auxiliary examination: Chest CT for assessment of lung infection

Chinese medicine treatments Chinese medicine treatments include oral administration of concentrated Chinese herbal decoction, fumigation/inhalation of Chinese medicine and vitamin C, and bolus administration of vitamin C.

Traditional Chinese and western medicine prescription details Traditional Chinese medicine treatment details Prescription 1: Buzhong Yiqi plus and minus formula (recommended for patients who had no fever and those who are in the convalescent period): This formula is composed of Radix Astragali 30 g, Radix Ginseng 15 g, Radix Glycyrrhizae 15 g, Rhizoma Atractylodis Macrocephalae 10 g, Pericarpium Citri Reticulatae 6 g, Radix Angelicae Sinensis 10 g, Fructus Jujubae 6, Rhizoma Zingiberis Recens 9 pieces, Radix Bupleuri 12 g, Rhizoma Cimicifugae 6 g.

Preparation method: The aforementioned herbs are decocted with water. After removal of macromolecules, 50 g concentrate is left, and then packaged, 25 g/dose.

Suggested usage: 1 dose once, twice a day, taking with warm water.

Prescription 2: Huhuang Detoxicity Paste (recommended for patients who have no fever): This formula is composed of Rhizoma Coptidis 20 g, Radix Et Rhizoma Rhei 10 g, Rhizoma Atractylodis 10 g, Radix Asteris 10 g, Herba Houttuyniae 10 g, Herba Taraxaci 10 g, Rhizoma Polygoni Cuspidati 10 g, Radix Astragali 20 g.

Preparation method: The aforementioned herbs are boiled with water. The extract was subjected to high-speed centrifugation. After removal of impurities, 50 g concentrate is left, and then packaged, 25 g/dose.

Suggested usage: One dose once, twice a day, taking with warm water.

Prescription 3: Baimu Qingre Jiedu Paste This formula is composed of Radix Puerariae 15 g, Radix Angelicae Dahuricae 12 g, Flos Magnoliae 9 g, Radix Isatidis 30 g, Fructus Forsythiae 15 g, Bulbus Fritillariae Thunbergii 12 g Preparation method: The aforementioned herbs are boiled with water. The extract was subjected to high-speed centrifugation. After removal of impurities, 50 g concentrate is left, and then packaged, 25 g/dose.

Suggested usage: One dose once, twice a day, taking with warm water.

Prescription 4: Fumigation/inhalation of Chinese herbs and vitamin C The formula consists of Rhizoma Coptidis 20 g, Radix Et Rhizoma Rhei 10 g, Rhizoma Atractylodis Macrocephalae 10 g, Radix Astragali 10 g, Radix Asteris 10 g, Herba Houttuyniae 10 g, Herba Taraxaci 10 g, Rhizoma Polygoni Cuspidati 10 g, Radix Astragali 20 g.

Preparation method: The aforementioned herbs are boiled with water. The extract was subjected to high-speed centrifugation. After removal of impurities, 50 g concentrate is left, and then packaged, 25 g/dose.

Fumigation/inhalation method: 3L of water is added to the intelligent rice cooker (specification 5L), and then the aforementioned semifluid paste is also placed in the cooker. After boiling, 10 g vitamin C is added. The oxygen tube is inserted into the bottom of the traditional Chinese medicine solution (oxygen flow is about 3-4 L/min). The steam is sucked with the mouth and nose alternately, 30-40 minutes once, 3-7 times a day. Patients take vitamin E capsule and folic acid every day.

Bolus administration of vitamin C 100 mL of 5% glucose containing vitamin C (10 g/60 kg body mass) is intravenously administered twice a day.

Western medicine treatment details Atomized inhalation of 5 million U α-interferon and 2 mL sterilized water, twice a day; 0.2 g arbidol, three times a day, treatment course no more than 10 days; intravenous administration of ribavirin 500 mg, once every 12 hours, treatment course no more than 10 days; intravenous administration of 10 g immunoglobulin C, once a day, 3-5 days. Anti-bacterial infection treatment is given to the patients who have yellow sputum and increased levels of procalcitonin and other bacterial infection specific indicators.

Notes for case and course record The medical record of integrated Chinese and western medicine treatment for each case should be carefully filled. A summary of the medical record is made every three days. The name and dosage of the traditional Chinese medicine and western medicine used, the route of administration, curative effect, and side effects are recorded. The record form of the curative effect should be filled every day.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mild and severe COVID-19 confirmed according to the Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial Version 7) that was issued by the National Health Commission & State Administration of Traditional Chinese Medicine;
2. Patients with suspected COVID-19 who meet one of the following pathogenic or serological evidence are also confirmed infected with the virus: a) COVID-19 nucleic acid test positive, as confirmed by real-time fluorescence RT-PCR detection; b) viral gene sequencing is highly homologous with the known COVID-19; c) serum test positive for both COVID-19 specific IgM and IgG antibodies; d) serum IgG antibody turns positive from negative or IgG antibody level in the recovering phase rises four times or higher than in the acute phase
3. Patients with moderate COVID-19 have fever and respiratory symptoms and present with the imaging features of coronavirus disease
4. Subjects will be considered developing severe COVID-19 if one of the following conditions occur: a) dyspnea, respiratory ≥ 30 beats/minute, blood oxygen saturation ≤ 93%, partial pressure of arterial oxygen (PaO2)/ fraction of inspired oxygen ratio (FiO2) ≤ 300, and /or lung infiltrates > 50% within 24 to 48 hours
5. Age > 18 years, of either sex Provision of written informed consent

Exclusion Criteria:

1. Patients with critical COVID-19 presenting with shock, acute respiratory distress syndrome, multiple organ failure
2. Patients with mild COVID-19
3. Pregnant or lactating woman
4. Upon the investigator's judgment, patients had the diseases that possibly influence patient participation in this study or study outcomes (such as malignant disease, autoimmune disease, severe malnutrition, liver and kidney disease, blood disease, nervous system disease, endocrine diseases) or currently suffer from the diseases that seriously affect the immune system (such as human immunodeficiency virus infection) or blood system, or splenectomy/organ transplantation.
5. Upon the request of the investigators or sponsors, patients with other acute malignant or chronic disease or mental disorder are not suitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Recovery time | From date of randomization until the date of discharge, assessed up to 6 months
  The discharge criteria of Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial Version 7) are applied: a) body temperature is back to normal for more than three days; b) respiratory symptoms improve obviously; c) pulmonary imaging shows obvious resolution of inflammation; d) nuclei acid tests negative twice consecutively on respiratory tract samples such as sputum and nasopharyngeal swabs (sampling interval being at least 24 hours)

SECONDARY OUTCOMES:
Time of disappearance of fever symptoms | From date of randomization until the date of discharge, assessed up to 6 months
  Time of disappearance of fever in degrees centigrade
The rate of conversion from COVID-19 positive to COVID-19 negative | From date of randomization until the date of discharge, assessed up to 6 months.
  The rate of conversion from COVID-19 positive to COVID-19 negative
Time of disappearance of cough | From date of randomization until the date of discharge, assessed up to 6 months
  Time of disappearance of cough in times per day
Respiratory rate | 1-14 days after treatment
  Respiratory rate in times/minute with blood gas analysis
Blood oxygen saturation | 1-14 days after treatment
  Blood oxygen saturation in percent with blood gas analysis
PaO2 | 1-14 days after treatment
  PaO2 in kPa with blood gas analysis
PaCO2 | 1-14 days after treatment
  PaCO2 in kPa with blood gas analysis
The time of obvious improvement as shown on chest CT scans relative to admission | From date of randomization until the date of discharge, assessed up to 6 months
  The time in days of patients of obvious improvement as shown on chest CT scans relative to admission
The rate of obvious improvement as shown on chest CT scans relative to admission | From date of randomization until the date of discharge, assessed up to 6 months
  The rate in percentages of patients of obvious improvement as shown on chest CT scans relative to admission
Levels of C-reactive protein | 1-14 days after treatment
  Levels of C-reactive protein measurement in mg/L
Erythrocyte sedimentation rate | 1-14 days after treatment
  Erythrocyte sedimentation rate in mm/h
Levels of Procalcitonin | 1-14 days after treatment
  Levels of Procalcitonin in ng/mL
Levels of interleukin-6 | 1-14 days after treatment
  Serum Levels of interleukin-6 in ng/L
Levels of interleukin-10 | 1-14 days after treatment
  Levels of interleukin-10 in ng/L
Levels of tumor necrosis factor-alpha | 1-14 days after treatment
  Levels of tumor necrosis factor-alpha in ng/mL

OTHER OUTCOMES:
Ultrasound examination of the urinary system | 1-14 days after treatment
  Ultrasound examination of the kidney, ureter, and bladder after treatment to mainly check for urolithiasis

CONTACTS AND LOCATIONS:
Overall Officials: Xijing He, MD, Study Chair — Xi'an International Medical Center Hospital; Yongping Liu, Principal Investigator — Xi'an International Medical Center Hospital; Xudong Yang, Principal Investigator — Xi'an International Medical Center Hospital; Yali Wang, Principal Investigator — Xi'an International Medical Center Hospital; Yifan Feng, Principal Investigator — Xi'an International Medical Center Hospital; Kuiwei Zhang, Principal Investigator — Xi'an International Medical Center Hospital; Jiayue Shan, Principal Investigator — Xi'an International Medical Center Hospital; Lei Shang, Principal Investigator — Xi'an International Medical Center Hospital; Zhijian Cheng, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University; Rui Wang, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University; Guoyu Wang, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University; Hui Gao, Principal Investigator — Xi'an International Medical Center Hospital; Shanjiao Jiang, Principal Investigator — Xi'an International Medical Center Hospital; Shenhao Liu, Principal Investigator — Xi'an International Medical Center Hospital
Locations (1):
- Xi'an International Medical Center Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No